CLINICAL TRIAL: NCT03972124
Title: Cannabis for the Prophylactic Treatment of Migraine: a Randomized Double-Blind Placebo-Controlled Clinical Trial
Brief Title: Cannabis for the Prophylactic Treatment of Migraine
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Farnaz Amoozegar, MD, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB19-0889
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD 100 mg OD (Active Comparator): The lower dose CBD group will start with CBD capsules 10 mg OD, then increase the dose every 4 days until on the target dose of 100 mg OD.
  Interventions: Drug: CBD 100 mg OD
- CBD 200 mg OD (Experimental): The higher dose CBD group will start with CBD capsules 10 mg OD and will increase every 4 days until on a target dose of 200 mg OD.
  Interventions: Drug: CBD 200 mg OD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD 100 mg OD — CBD oil - purified to <1% THC in soft-gel capsules
  Arms: CBD 100 mg OD
Drug: CBD 200 mg OD — CBD oil - purified to <1% THC in soft-gel capsules
  Arms: CBD 200 mg OD
Drug: Placebo — Soft-gel capsules containing placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of cannabis for the treatment of chronic migraine headaches. Study subjects will be randomized to one of three groups: lower dose CBD, higher dose CBD or placebo.

DETAILED DESCRIPTION:
Migraine is a neurological disorder characterized by recurrent attacks of moderate to severe headache, often accompanied by sensory sensitivity and nausea. Migraine can be very disabling and often interferes with social and occupational functioning.

Given the high prevalence of migraine and the significant burden it places on the individual and society, it is an important condition to study and manage optimally. This is especially true because current migraine treatments often result in only marginal improvement and are frequently associated with intolerable side effects. For this reason, there is a need for new migraine treatments. The endocannabinoid system is an important potential treatment target as it is involved in pain processing and overlaps with some mechanisms of migraine pathophysiology.

Cannabis was legalized in Canada on October 17th, 2018. As a result, the consumption of cannabis products for migraine treatment may increase. However, at this time there is limited evidence for the safety and efficacy of cannabis for the treatment of migraine. As a result, there is a need for further study and research in this area. Thus, we propose a randomized, double-blind, placebo-controlled clinical trial to study cannabis (specifically cannabidiol) as a preventative therapy for patients with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give signed informed consent.
* Male and female patients aged 25 years or older.
* History of migraine for at least 12 months as diagnosed by the International Classification of Headache Disorders (ICHD-3).
* Chronic migraine for at least the previous 3 months prior to screening, as diagnosed by ICHD-3.
* Migraine preventative medications (including Botulinum toxin injections) are permitted if dose is stable for the 3 month period prior to randomization, and no change to dose is planned for the entire duration of the study.
* Using a reliable method of contraception for females of child-bearing age.
* Failure of at least 2 prior migraine preventatives, either due to lack of efficacy with an appropriate trial of the medication, or due to lack of tolerability.
* Able to follow study procedures, fill out headache diaries, and complete questionnaires.
* Completion of at least 90% of the headache diary during the one month baseline period.

Exclusion Criteria:

* Other active primary headaches, such as cluster headache, hemicrania continua, etc.
* Any secondary headache, such as headache related to intracranial hypertension, intracranial hypotension, hydrocephalus, intracranial mass lesion, etc.
* Pregnant, planning to become pregnant, or breastfeeding.
* Active or significant history of major mental illness, including severe depression, or anxiety, and any history of psychosis or schizophrenia.
* History of or current substance use disorder.
* Regular use of cannabis for medical or recreational reasons during the previous 12 months.
* History of significant cardiovascular or cerebrovascular disease, such as previous myocardial infarction, stroke, or peripheral vascular disease.
* History of hypertension greater than 160/100 and not medically treated.
* Any past history of seizure disorder.
* Liver disease or liver enzymes two or more times the upper limit of normal at baseline.
* Severe renal disease or GFR more than 30% below expected.
* Any disorder or condition leading to hypersomnolence or excessive daytime drowsiness, such as narcolepsy, excessive use of sedatives/hypnotics, etc.
* Any other medical condition that in the opinion of the investigators may pose a health risk to the subject if entered into the clinical trial.
* Use of interventions or devices, such as nerve blocks, sphenopalatine ganglion blocks, vagal nerve stimulators, and transcranial magnetic stimulators during the baseline period (weeks -4 to 0). These treatments will also be prohibited during the period of therapy (weeks 0 to 12).
* Use of transitional therapies such as a course of steroids or a dihydroergotamine protocol during the baseline period (weeks -4 to 0). These treatments will also be prohibited during the period of therapy (weeks 0 to 12).
* Overuse of triptan, dihydroergotamine, opioid, or barbiturate medications, defined as 10 or more days per month in the 3 months prior to randomization.
* Overuse of simple analgesics (such as acetaminophen, ibuprofen, aspirin), and non-steroidal anti-inflammatories (such as naproxen, ketorolac, diclofenac, etc.) defined as 15 or more days per month in the 3 months prior to randomization.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The mean change in the number of headache days between the 4-week baseline period compared to the 4-week period just preceding the 3 month follow-up visit. | Baseline and weeks 9-12

SECONDARY OUTCOMES:
The mean change in the number of headache days between baseline compared to the 4-week period just preceding the 6 month follow-up visit. | Weeks -4 to 0 and weeks 21-24
The percentage of patients who have at least a 50% reduction in their headache frequency between baseline compared to weeks 9-12 (the 50% responder rate). | Weeks -4 to 0 and weeks 9-12
The change in the mean headache intensity between baseline compared to weeks 9-12, and weeks 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
The mean change in the number of days with acute pain medication use between baseline compared to weeks 9-12, and 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
Change in Migraine Disability Assessment (MIDAS) Test score between baseline compared to weeks 9-12, and 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
  The MIDAS test assesses the impact of migraines on daily life. The score ranges between 0 and 21+ with a lower score indicating little or no disability and a higher score indicating severe disability.
Change in Headache Impact Test (HIT-6) score between baseline compared to weeks 9-12, and 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
  The HIT-6 test score ranges between 36-78 with a higher score being associated with greater impact of headache on an individual's life.
Change in Generalized Anxiety Disorder (GAD-7) score between baseline compared to weeks 9-12, and 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
  The GAD-7 patient questionnaire is used as a screening tool for generalized anxiety disorder with scores ranging between 0-21. A higher score is associated with a probable diagnosis of severe anxiety.
Change in Patient Health Questionnaire (PHQ-9) score between baseline compared to weeks 9-12, and 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
  The PHQ-9 questionnaire is a self-administered screening tool for depression. The questionnaire score can range between 0-27 with higher scores indicating severe depression.
Change in Migraine Specific Quality of Life Questionnaire (MSQ) score between baseline compared to weeks 9-12, and 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
  The MSQ assesses the impact (restrictive, preventative and emotional) of migraine on an individual's quality of life.
Change in the Pittsburgh Sleep Quality Index (PSQI) score between baseline compared to weeks 9-12, and 21-24. | Weeks -4 to 0, weeks 9-12 and weeks 21-24
  The PSQI is a tool used to measure the quality of an individual's sleep. The PSQI is self-administered with a higher score indicating overall poor sleep.